CLINICAL TRIAL: NCT05883098
Title: Effectiveness of Supra SDRM® vs. Fibracol Plus Collagen in the Treatment of Diabetic Foot Ulcers: a Pilot Randomized Controlled Trial
Brief Title: SDRM® vs. Collagen for Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polymedics Innovations Inc. (Industry)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMI-SUPRASDRM®-01
Record Dates: First submitted 2023-05-08; First posted 2023-05-31 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot; Ulcer Foot; Wound Heal
Keywords: Diabetic foot ucer; Wound closure matrix; Wound healing; Chronic wound
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SUPRA SDRM (Experimental): The subject will receive wound standard of care that will include Supra SDRM as an active synthetic wound closure matrix, covered with a non-adherent dressing plus an appropriate outer dressing to maintain moisture balance, then wrapped with stretch gauze and self-adherent wrap. Supra SDRM will be applied weekly, and the exterior dressings will be redressed as necessary.
  Supra SDRM is FDA-cleared (K090160, K170213) for the management of partial and full-thickness wounds, such as pressure sores, leg ulcers, diabetic ulcers, and surgical wounds. It is commercialized as a single dermal substitute matrix for wound management. No preparation of SUPRA SDRM matrix is necessary. When applied to the wound SUPRA SDRM adheres well to the wound bed without the need for direct fixation. SUPRA SDRM becomes translucent after the application allowing healthcare professionals to easily assess the wound healing. SUPRA SDRM® is available in multiple sizes and can be trimmed to meet the patient's needs.
  Interventions: Procedure: Wound debridement; Device: Wound closure matrix application
- Fibracol Plus (Active Comparator): The subject will receive wound standard of care that will include Fibracol Plus collagen dressing as an active synthetic wound closure matrix, covered with a non-adherent dressing plus an appropriate outer dressing to maintain moisture balance, then wrapped with stretch gauze and self-adherent wrap. Fibracol Plus collagen dressing will be applied weekly, and the exterior dressings will be redressed as necessary.
  FIBRACOL™ Plus Collagen Wound Dressing with Alginate dressing contains more than just pure collagen. It's a soft, absorbent, and conformable wound dressing, composed of 90% collagen and 10% calcium alginate. In the presence of wound fluid, FIBRACOL™ Plus Dressing helps maintain a physiologically moist microenvironment at the wound surface. This environment supports granulation tissue formation, epithelialization and rapid wound healing.
  Interventions: Procedure: Wound debridement; Device: Wound closure matrix application

INTERVENTIONS:
Procedure: Wound debridement — The study's wounds will be mechanically debrided before the experimental or active comparator devices are applied. Debridation will be performed by a trained clinician using a curette. Necrotic tissue and slough will be removed during this procedure.
Device: Wound closure matrix application — After wound debridement, the patients will receive the application of a wound closure matrix as dictated by their randomization allocation.

SUMMARY:
Supra SDRM® is FDA-cleared as a dressing for treating partial and full-thickness wounds. It is a dermal substitute that provides a barrier and an ECM-like structure to help accelerate wound healing. SUPRA SDRM® has 510k approval for partial and full-thickness wounds and has shown promising results in preliminary animal studies. The purpose of this clinical evaluation is to collect and compare outcomes data from patients with UT 1A diabetic foot ulcers treated with a commercially available dermal substitute, Supra SDRM®, as compared to an advanced standard of care (Fibracol Plus). Patient outcomes, including time to heal, healing by 12 weeks, direct costs, and infection rate, will be compared at the end of the study.

DETAILED DESCRIPTION:
Chronic wounds are those that fail to proceed through the normal phases of wound healing. They pose a high risk for infection and risk complications resulting in amputation. A plethora of wound treatment modalities are commercially available to help improve patient outcomes. However, even when combined with a good standard of care practices and wound dressings, they may not be sufficient to promote timely wound closure. Cellular and/or tissue- based products (CTPs) may provide a healing advantage over traditional dressings. CTPs are derived from human (allograft), animal (xenograft), or synthetic materials or a combination thereof. CTPs can help encourage tissue repair or regeneration by providing scaffolds and the cells necessary to stimulate wound healing. Synthetic products may provide advantages over human or other animal sourced products because they are natural, non-biologic, avoid complications due to risk of disease transmission, and possess less immunologic potential.

The fully synthetic skin substitute evaluated in this study is SUPRA SDRM® Synthetic Biodegradable Matrix Wound Dressing (Polymedics Innovations Inc.; Woodstock,GA). The device is a novel synthetic, guided wound closure matrix, built as a bimodal foam membrane structure for the management of chronic wounds. It combines the benefits of a microporous structure that builds a protective barrier allowing the wound to heal and additional large pores which were created to enable ingrowth of blood vessels. This microenvironment initially provides a seal against contamination and modulates inflammation in wound bed. Subsequently, it supports cellular processes required for tissue repair and wound healing.

In this parallel randomized clinical trial, patients with diabetic foot ulcers grade UT 1A will receive either standard of care plus SUPRA SDRM or a collagen dressing (Fibracol Plus) weekly after wound debridement. Primary outcomes will be time to achieve wound healing, and the proportion of patients achieving healing by 12 weeks. Secondary outcomes will include the direct costs of treatment and the proportion of patients who developed infections during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 or older.
* Subject is willing to sign an informed consent and participate in all procedures and follow-up evaluations.
* Study ulcer is diabetic in origin, located on foot or below the malleolus (UT Grade 1A).
* Study ulcer size is a minimum of 2 cm2 and a maximum of 25 cm2.
* Study ulcer has been present for a minimum of 4 weeks before enrollment and less than 1 year old.
* Study ulcer has been offloaded for at least 14 days before randomization.
* Subject does not exhibit clinical signs or symptoms of infection.
* Subject has adequate control of diabetes demonstrated by Hemoglobin A1c < 12% within 90 days of screening.
* Subject has adequate circulation to the affected extremity.

Exclusion Criteria:

* Study ulcer has > 40% wound healing during the 14 days screening period.
* Subject has a known history of poor compliance with medical treatments.
* Subject is presently participating in another clinical trial.
* Subject has a known or suspected local or systemic malignancy.
* Subject has been diagnosed with autoimmune connective tissues diseases.
* Subject has received graft material or topical growth factors on the study ulcer within the previous 30 days.
* Subject has received application of topical steroids on the study ulcer surface within the previous 30 days.
* Subject is pregnant or breast feeding.
* Subject is on dialysis.
* Subject is taking medications that are considered immune system modulators or cytotoxic chemotherapies.
* Subject cannot be on systemic antibiotics prior to randomization, however, during the treatment phase infection management may include systemic antibiotics if in conjunction with debridement.
* Subject has a known allergy to ingredients/components of Supra SDRM®.
* Subject has osteomyelitis, and/or bony prominences present in the wound.
* Subject has ulcer probing to bone and tendon. (UT Grade II or III A-D).
* Subject is unable to comply with planned study procedures and treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Time to heal | Up to 30 weeks
  Number of weeks required to achieve 100% epithelization of the wound
Healing by 12 weeks | 12 weeks
  Proportion of patients achieving 100% epithelization on or before week 12

SECONDARY OUTCOMES:
Direct costs | Up to 30 weeks
  Direct costs of treatment
Infection rate | Up to 30 weeks
  Proportion of patients developing an infection in the wound bed

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Ramirez Garcia Luna, MD, PhD, Study Chair — McGill University; Brock A Liden, DPM, Principal Investigator — WAFL Inc
Locations (1):
- WAFL Inc, Circleville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frykberg RG, Banks J. Challenges in the Treatment of Chronic Wounds. Adv Wound Care (New Rochelle). 2015 Sep 1;4(9):560-582. doi: 10.1089/wound.2015.0635. PMID 26339534
- [Background] Mirhaj M, Labbaf S, Tavakoli M, Seifalian AM. Emerging treatment strategies in wound care. Int Wound J. 2022 Nov;19(7):1934-1954. doi: 10.1111/iwj.13786. Epub 2022 Mar 17. PMID 35297170
- [Background] Haller HL, Sander F, Popp D, Rapp M, Hartmann B, Demircan M, Nischwitz SP, Kamolz LP. Oxygen, pH, Lactate, and Metabolism-How Old Knowledge and New Insights Might Be Combined for New Wound Treatment. Medicina (Kaunas). 2021 Nov 1;57(11):1190. doi: 10.3390/medicina57111190. PMID 34833408